CLINICAL TRIAL: NCT06867198
Title: Impact of Peanuts on Cardiometabolic, Cognitive, and Intestinal Health in Prediabetes Among Racially Diverse Populations
Brief Title: Peanuts for Cardiometabolic, Brain, and Intestinal Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); The Peanut Institute (Other)
Responsible Party: Principal Investigator, Rafaela G. Feresin, Associate Professor, Georgia State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H25014
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prediabetes; Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Cognition; Microvascular Function; Gut Microbiota; Endothelial Function (Reactive Hyperemia); Arterial Stiffness, Blood Pressure; Adult
Keywords: prediabetes; peanuts; functional foods; nuts; metabolic health; insulin resistance; type II diabetes; microvascular function; dietary intervention; cognitive function; vascular function; neuroimaging; endothelial function; cardiovascular health; gut microbiota
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance; Hyperemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peanut (Experimental): 43 g of peanut butter (1snack cup) 3 x/week, 42 g of dry roasted peanuts (1/3 of a cup) 3x/week, or 56 g of peanut flour 1x/week for 6 months
  Interventions: Dietary Supplement: Peanuts
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Peanuts — 43 g of peanut butter (1 snack cup) 3 x/week, 42 g of dry roasted peanuts (1/3 of a cup) 3x/week, or 56 g of peanut flour 1x/week for 6 months.
  Arms: Peanut

SUMMARY:
The overall objective of this 13-month randomized crossover study is to seek evidence demonstrating that daily consumption of peanuts and peanut products improve cardiometabolic, cognitive, and intestinal health in a racially diverse prediabetes population.

DETAILED DESCRIPTION:
In the US, 37.1 million adults have diabetes mellitus and 96 million have prediabetes. Type 2 diabetes mellitus (T2DM) accounts for 95% of the cases and results in many public health complications that increase economic burden and reduce productivity and quality of life. Eight out of 10 people with T2DM die from cardiovascular disease, while those with T2DM also face a 50% higher risk of developing dementia compared to healthy individuals. Also, studies indicate that intestinal health significantly influences the development of T2DM. Of note, the burden of T2DM is particularly pronounced in non-Hispanic Black and Hispanic populations compared to the non-Hispanic White population. Prevention and treatment of T2DM focus on lifestyle changes including dietary modifications. Plant-based foods, including peanuts and peanut products, have been increasingly recognized for their importance in the prevention and management of prediabetes and T2DM due to their unique nutritional profile, including their favorable fatty acid composition, fiber content, and bioactive compounds. While emerging evidence indicates that peanut improves cardiometabolic, cognitive and intestinal health, no studies have collectively and comprehensively evaluated the effects of peanut or peanut product consumption on the cardiometabolic, cognitive, and intestinal health of individuals with prediabetes or T2DM. Thus, this study aims to investigate whether adults with prediabetes consuming 43 g of peanut butter (1 snack cup) 3 x/week, 42 g of dry roasted peanuts (1/3 of a cup) 3x/week, or 56 g of peanut flour 1x/week for six months will have 1) reduced levels of serum HbA1c, fasting glucose (FBG), insulin, HOMA-IR (homeostatic model assessment of insulin resistance) and improved lipid profile, 2) reduced blood pressure, improved endothelial function, arterial stiffness and microvascular function, 3) Improved gut microbiota composition and reduced intestinal permeability, 4) improved cognitive function (verbal memory and executive functions [inhibition, working memory, cognitive flexibility]) and brain health metrics as assessed by neuroimaging, and 5) reduced serum markers of oxidative stress and inflammation. The effectiveness of the intervention on the abovementioned outcomes among races including non-Hispanic Black (NHBA), non-Hispanic White (NHWA), non-Hispanic Asian (NHAA) and Hispanic (HA) adults will also be compared. Lastly, whether changes in cardiometabolic and cognitive outcomes are associated with changes in intestinal microbiota outcomes and whether changes in cardiometabolic outcomes are associated with changes in cognitive function parameters will be explored.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 20-59 years of age
* Prediabetes (fasting blood glucose levels 100-125 mg/dL and/or HbA1c between 5.7-6.4%)

Exclusion Criteria:

* Allergies to peanuts and peanut products
* Use of insulin, antidiabetic, antibiotics, and anti-inflammatory drugs
* Active cancer, gastrointestinal, renal, cardiovascular, thyroid, and neurological diseases or severe head injury
* Smoking
* Consumes greater than 2 alcoholic beverages per day
* Consumes antioxidant, probiotic, and prebiotic supplements
* Pregnant or Lactating
* Actively participating in a weight loss program

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | Baseline, 3 months, and 6 months
  Measurement of fasting blood glucose
Glycosylated hemoglobin | Baseline, 3 months, and 6 months
  Measurement of fasting glycosylated hemoglobin

SECONDARY OUTCOMES:
Ambulatory Blood Pressure | Baseline, 3 months, and 6 months
  Assessment of whole-day ambulatory blood pressure during daytime and nighttime periods.
Fasting Insulin | Baseline, 3 months, and 6 months
  Measurement of fasting insulin
Homeostasis model assessment-insulin resistance (HOMA-R) | Baseline, 3 months, and 6 months
  Calculated as fasting insulin (mU/mL) x fasting glucose (mg/dL)/405
Blood Lipid Profile | Baseline, 3 months, and 6 months
  Measurement of blood lipid profile
Gut Microbiota Composition | Baseline, 3 months, and 6 months
  Analysis of stool sample for determination of absolute levels of bacteria and relative species composition
Global Cognitive Ability | Baseline, 3 months, and 6 months
  Measured using NIH Toolbox Picture Vocabulary test and Oral Reading Recognition
Performance Validity | Baseline, 3 months, and 6 months
  Assessed using Rey 15
Verbal Memory & Recognition | Baseline, 3 months, and 6 months
  Measured using Rey Auditory Verbal Learning Test with appropriate alternate forms
Cognitive Inhibition | Baseline, 3 months, and 6 months
  Measured using Delis-Kaplan Executive Function System Color Word Interference, and NIH Toolbox Flanker Inhibitory Control and Attention
Cognitive Flexibility | Baseline, 3 months, and 6 months
  Assessed using Delis-Kaplan Executive Function System Trails and Verbal Fluency Switching
Working Memory | Baseline, 3 months, and 6 months
  Measured using Digit Span and NIH Toolbox List Sorting
Processing Speed | Baseline, 3 months, and 6 months
  Measured using NIH Toolbox Pattern Comparison and Oral Symbol Digit tests
Associative Memory | Baseline, 3 months, and 6 months
  Measured using NIH Toolbox Face Name Associative Memory Exam and Face Name Associative Memory Exam Delay tests
Attention | Baseline, 3 months, and 6 months
  Assessed using Wechsler Adult Intelligence Scale - IV and Rey Auditory Verbal Learning Test Trial 1
Problem-Solving | Baseline, 3 months, and 6 months
  Assessed using NIH Toolbox Visual Reasoning Test

OTHER OUTCOMES:
Reactive Hyperemia Index | Baseline, 3 months, and 6 months
  Assessment of endothelial function in response to increased shear stress using EndoPAT2000
Pulse Wave Velocity | Baseline, 3 months, and 6 months
  Arterial Stiffness will be assessed by pulse wave velocity using SphygmCor
Percent Maximal Microvascular Blood Flow | Baseline, 3 months, and 6 months
  Micro-vessel blood flow in response to local heating stimulus will be assessed using a Laser Doppler
Circulating Markers of Inflammation and Oxidative Stress | Baseline, 3 months, and 6 months
  Measurement of concentrations of circulating markers of inflammation such as CRP and oxidative stress such as TBARS in blood plasma and serum samples
Urinary Polyphenolic Metabolites | Baseline, 3 months, and 6 months
  24-hour urine collection samples will be assessed for polyphenol metabolites
Body Fat | Baseline, 3 months, and 6 months
  DEXA will be used to assess body fat.
Spontaneous brain activity at rest | Baseline and 6 months
  Assessed with resting state-functional Magnetic Resonance Imaging
Blood flow (perfusion) in the brain | Baseline and 6 months
  Assessed with Arterial Spin Labeling Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela G Feresin, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States